CLINICAL TRIAL: NCT07125040
Title: Characterization of the Natural History of Laminin-Alpha-2-Related Dystrophy (LAMA2-RD) Patients and Identification of Novel Disease Biomarkers
Brief Title: Characterization of the Natural History of LAMA2-RD and Identification of Novel Disease Biomarkers
Status: Recruiting | Type: Observational
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Alberto Andrea Zambon, MD, PhD - Principal Investigator, Università Vita-Salute San Raffaele
Other Study IDs: GUP24002_LAMA2
Record Dates: First submitted 2025-07-17; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: LAMA2-MD (Merosin Deficient Congenital Muscular Dystrophy, MDC1A); LAMA2-MD (Merosin Deficient Congenital Muscular Dystrophy, MDC1A); Merosin Deficient CMD (Full or Partial); Merosin Deficient Congenital Muscular Dystrophy
Keywords: LAMA2-RD; Natural history
MeSH Terms: conditions — Muscular dystrophy congenital, merosin negative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cardiac MRI — On a subset of adult patients

SUMMARY:
The goal of this observational study is to learn about the natural history and multi-organ involvement of Laminin-Alpha-2-Related Dystrophy (LAMA2-RD) in pediatric and adult patients. The main questions it aims to answer are:

* What is the prevalence and nature of cardiac involvement, and how do this relate to age and muscular phenotype?
* What is the prevalence of peripheral neuropathy, and how do this relate to age and muscular phenotype?
* What is the extent of respiratory, nutritional, skeletal, and cognitive/brain involvement, particularly in adults with more severe vs less severe phenotypes?
* How does quality of life and transition to adulthood occur in individuals with LAMA2-RD?
* Which nomenclature best reflects differences in disease severity and may support future clinical trial design?

Study participants will:

* Undergo retrospective and prospective clinical assessments every 12 months for 2 years across multiple centers.
* A subset of adult participants (n=20) will receive cardiac MRI with contrast enhancement.
* Provide biological samples during routine blood testing for future research.

DETAILED DESCRIPTION:
Background: LAMA2-RD is an autosomal recessive disorder due mutations in the LAMA2 gene. The clinical manifestations of LAMA2-RD range from severe, early-onset congenital muscular dystrophy (CMD) to a milder limb-girdle type muscular dystrophy (LGMDR23). A few promising therapies are getting closer to clinical application, but clinical trial readiness is limited by the paucity of natural history studies. Although some groups have recently shed light on different aspects of the disease, these are usually focused on pediatric populations. A detailed description of the disease in adult patients as well as the importance of specific organs involvement (e.g., heart and peripheral nervous system) are lacking.

Objectives: To describe the natural history of a large cohort of patients affected by LAMA2-RD (n=40-45).

Specifically, the investigators aim 1) to clarify the prevalence and characteristics of cardiac involvement, and to correlate the latter with age and muscular phenotype 2) to clarify the degree of neuropathic involvement 3) to clarify respiratory, nutritional, skeletal, and brain/cognitive involvement, with a focus on adult population 4) to clarify which nomenclature better captures differences in terms of disease severity, to help refine inclusion criteria for trials 5) to understand how quality of life is impacted and transition to adulthood performed 6) to collect biological material for future research Design and methods: This will be a multicenter, retrospective and prospective longitudinal observational study with additional procedures for a subset of patients: cardiac MRI with contrast enhancement and an additional sample handling during routine blood test. Patients will be assessed every 12 months over a period of 2 years. In addition to routine clinical assessments, cardiac MRI will be performed in a selected 20 adult population. The differential involvement of specific organs between LAMA2-RD subpopulations will be analyzed.

ELIGIBILITY:
INCLUSION

Diagnosis of LAMA2-related dystrophy confirmed via:

1. Two causative mutations in the LAMA2 gene or Muscle biopsy with absence of
2. merosin (laminin-211) and at least one causative mutation in the LAMA2 gene or

   * Consistent phenotype and affected siblings with criteria a) or b) and
   * Ability to participate in study visits at least every 12 months during a 24 months period.
   * Ability to sign informed consent for adults or parents/ legal tutors for children

EXCLUSION

* Lack of a confirmed diagnosis of LAMA2-relate dystrophy
* Inability to participate in study visits at least every 12 months
* Medical fragility which precludes the ability to safely travel to the study site and/or participate in the study assessments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric patients affected by LAMA2-RD
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Rhythm abnormalities | 0, 12, 24 months
  Prsence or absence of rhythm abnormalities (Brady arrhythmia, supraventricular and ventricular tachyarrhythmia) as detected by ECG and 24-hour Holter ECG
Cardiac function | 0, 12, 24 months
  Left ventricular end-diastolic volume (LVEDV) and left ventricular ejection fraction (LVEF) measured by transthoracic echocardiogram
Cardiac inflammation and fibrosis | T0
  Cardiac inflammation and fibrosis by cardiac Magnetic Resonance Imaging (MRI) (only in adult patients)

SECONDARY OUTCOMES:
Motor outcome 1 | 0, 12, 24 months
  The Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND) (0-2 years); maximum score 64
Motor outcome 2 | 0,12, 24 months
  Motor Function Measure (MFM20 2-5 years; maximum score 60; MFM32 ≥ 5 years; maximum score 96)
Motor outcome 3 (Upper limbs) | 0, 12, 24 months
  Upper limbs function: Performance upper limb module 2.0. (PUL 2.0); maximum score 42
Motor outcome 4 (Timed tests) | 0, 12, 24 months
  6 minutes walk test (6MWT) - metres
Motor outcome 4 (Timed tests) | 0, 12, 24 months
  Timed rise from the floor (TRF) - seconds
Motor outcome 5 | 0, 12, 24 months
  North Star Assessment for Limb-Girdle Type Muscular Dystrophies (NSAD); maximum score 54
Respiratory function | 0, 12, 24 months
  Lung function measurement (Forced vital capacity -FVC L/%predicted
Respiratory function | 0, 12, 24 months
  Forced Expiratory Volume in 1 second -- FEV1 L/%predicted
Respiratory function | 0, 12, 24 months
  Maximal Inspiratory Pressure- MIP
Respiratory function | 0, 12, 24 months
  Maximal Expiratory Pressure - MEP
Respiratory function | 0, 12, 24 months
  Peak exploratory flow - PEF
Respiratory function | 0, 12, 24 months
  Peak cough flow - PCF

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Ospedale San Raffaele, Milan, Italy